CLINICAL TRIAL: NCT04687683
Title: Comparison of Immediate Effects of Different Posterior Shoulder Stretching Techniques in Overhead Athletes With Glenohumeral Internal Rotation Deficits
Brief Title: Comparison of Immediate Effects of Different Shoulder Stretching Techniques in Overhead Athletes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Gonca Şahiner Pıçak, Principal Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5002-GOA
Record Dates: First submitted 2020-12-15; First posted 2020-12-29 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Glenohumeral Internal Rotation Deficit

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Post Isometric Relaxation Group (Experimental): The participants in this group will receive post isometric relaxation stretching in modified cross body position.
  Interventions: Other: Post Isometric Relaxation Group
- Isolytic Stretching Group (Experimental): The participants in this group will receive isolytic stretching in modified cross body position.
  Interventions: Other: Isolytic Stretching Group
- Static Stretching Group Group (Experimental): The participants in this group will receive static stretching in modified cross body position.
  Interventions: Other: Static Stretching Group Group

INTERVENTIONS:
Other: Post Isometric Relaxation Group — Athletes will be positioned in a modified cross-body position. They will be asked to actively bring their underlying arm in the direction of horizontal adduction up to the physiological barrier barrier. The participants will be asked to perform an isometric contraction for 5 seconds in the horizontal abduction direction with 20% of the maximum muscle strength. After the relaxation, the arm will be moved towards horizontal adduction and 15 seconds active-assistive stretching will be applied. Participants will be given a 5-second rest period between contractions. This stretching exercise will be applied in 5 repetitions for one session.
  Arms: Post Isometric Relaxation Group
Other: Isolytic Stretching Group — Athletes will be positioned in a modified cross-body position. They will be asked to actively bring their underlying arm in the direction of horizontal adduction up to the physiological barrier barrier. The participants will be asked to perform a contraction in the horizontal abduction direction with 20% of the maximum muscle strength. When the muscle contraction occurs, the arm will be moved quickly in 2-4 seconds towards horizontal adduction and 15 seconds active-assistive stretching will be applied. Participants will be given a 5-second rest period between stretches. This stretching exercise will be applied in 5 repetitions for one session.
  Arms: Isolytic Stretching Group
Other: Static Stretching Group Group — Athletes will be positioned in a modified cross-body position. They will be asked to actively bring their underlying arm in the direction of horizontal adduction up to the physiological barrier. Then, the arm will be moved towards horizontal adduction and 15 seconds active-assistive stretching will be applied. Participants will be given a 5-second rest period between stretching exercises. This stretching exercise will be applied in 5 repetitions for one session.
  Arms: Static Stretching Group Group

SUMMARY:
81 overhead athletes with Glenohumeral Internal Rotation Deficit (GIRD) will be included in this study. Participants will be randomly divided into 3 different groups of 26 people. In each group will be applied posterior shoulder stretching exercises (PSSE) performed with different Muscle Energy Techniques (MET).

DETAILED DESCRIPTION:
Post Isometric Relaxation Group (PIRG) participants will perform a PSSE with post isometric relaxation (PIR) technique, Isolytic Stretching Group (ISG) participants will perform a PSSE with isolytic stretching technique and Static Stretching Group Group (SSG) participants will perform a PSSE with static stretching technique. All exercises will be performed in the modified cross-body position. Subacromial space and posterior capsule thickness will be measured using a 7-12 MHz linear transducer with USG (LOGIQ e Ultrasound, GE Healthcare, USA). Athletes' GIRD results and rotational ROM measurements will be measured and recorded using a bubble inclinometer (Fabrication End Inc, New York, USA). The upper extremity functional performance of the athletes will be evaluated with the Functional Throwing Performance Index (FTPI). Evaluations will be repeated tree times before, after the stretching exercise and 30 minutes later and the effects of different muscle energy techniques (MET) will be compared. Investigators hypothesized PSSE made with different MET techniques have different effects on Acromio-Humeral Distance, posterior capsule thickness, rotational ROM measurements and performance on overhead athletes with GIRD and the effects of MET would be superior to static stretching.

ELIGIBILITY:
Inclusion Criteria:

* Being overhead athlete
* Glenohumeral internal rotation range of motion of the affected shoulder should be less than other shoulder and bilateral shoulder internal rotation range of motion difference should be ≥15 º

Exclusion Criteria:

* Shoulder pain required medical attention for the last year.
* Current shoulder pain
* Cervical pain during upper extremity movement
* History of fracture to the shoulder girdle
* Systemic musculoskeletal disease
* History of shoulder surgery,
* Glenohumeral instability (positive apprehension, relocation, or positive sulcus test) or positive findings for a full thickness rotator cuff tear (positive lag sign, positive drop arm test, or marked weakness with shoulder external rotation)

Ages: 13 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 81 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Shoulder internal rotation range of motion | baseline measurements, 3 minutes and 30 minutes
  Change of shoulder internal rotation range of motion (with bubble inclinometer)

SECONDARY OUTCOMES:
Subacromial space | baseline measurements, 3 minutes and 30 minutes
  Change of subacromial space ( with Ultrasound)
Posterior capsule thickness | baseline measurements, 3 minutes and 30 minutes
  Change of posterior capsule thickness ( with Ultrasound)
Functional Throwing Performance Index | baseline measurements, 3 minutes and 30 minutes
  Participants will throw a ball to shot a frame on a wall. Number of correct shots will be recorded
Shoulder Total rotation range of motion | baseline measurements, 3 minutes and 30 minutes
  Change of shoulder internal rotation + external rotation range of motion (with bubble inclinometer)
Posterior shoulder tightness | baseline measurements, 3 minutes and 30 minutes
  Change of posterior shoulder tightness (with bubble inclinometer)

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi Sevi Yeşilyaprak, Phd, Study Director — Dokuz Eylul University